CLINICAL TRIAL: NCT02648321
Title: Motivational Intervention of Exercise in Patients With Psychosis
Brief Title: Motivational Intervention for Physical Activity in Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 13-482
Record Dates: First submitted 2015-12-10; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Psychotic Disorders
Keywords: Motivational Interviewing; Exercise
MeSH Terms: conditions — Psychotic Disorders; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): Motivational Interviewing
  Interventions: Behavioral: Motivational Interviewing
- Health Education (Active Comparator): Health Education
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing is a patient-centered, tailored counselling intervention for exercise, through which patients' motives to change are identified. Personal ideas and ambivalence are explored. The discrepancies between the present behavior and the patient's own future goals are amplified. The patient's intrinsic motivation for change is increased through the process.
  Arms: Motivational Interviewing
Behavioral: Health Education — General education about healthy lifestyle and diet.
  Arms: Health Education

SUMMARY:
The purpose of this study is to determine whether motivational intervention is effective in promoting exercise habit in patients with psychosis.

DETAILED DESCRIPTION:
The current study aims to investigate the beneficial effect of motivational intervention in promoting exercise habit in patients with psychosis. Outpatients will be recruited and will be randomized to a 12-week motivational intervention program. They will be assessed for their clinical symptoms, cognitive function, physical fitness, and quality of life. All patients will have cognitive function assessments at baseline, 12 weeks after the completion of the program and 6 months. The primary hypothesis of the current study is that motivational intervention can help patient to develop exercise habit in patients with early psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed to have psychotic disorders
* Cantonese-speaking Chinese (to enable cognitive testing)
* Ability to understand the nature of the study and to give written informed consent

Exclusion Criteria:

* Severe physical illness (Myocardial Infarction, Hypertension, Fracture, Spinal problems in which exercise may be contraindicated), and seizure disorders
* Comorbid substance dependence
* Unstable psychotic symptoms
* Known pregnancy
* A history of brain trauma or organic brain disease
* Known history of intellectual disability or special school attendance

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | 12 weeks

SECONDARY OUTCOMES:
Role Functioning Scale | 12 weeks
Short Form 36 | 12 weeks
PANSS | 12 weeks
Physical Activity Level | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No